CLINICAL TRIAL: NCT03342599
Title: Effects of Alpha Lipoic Acid Supplementation on Metabolic Syndrome Markers in Young Overweight or Obese Males
Acronym: ALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Verne (Other)
Responsible Party: Principal Investigator, Dr. Sarah L. Dunn, Associate Professor of Kinesiology, University of La Verne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ULVALApilot-01; ULV2013-CASIRB-24 (Other: University of La Verne)
Record Dates: First submitted 2015-02-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Alpha Lipoic Acid
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GNC Alpha Lipoic Acid Supplement (Experimental): 600mg/daily ingestion of GNC alpha lipoic acid with no change in lifestyle for 8 weeks
  Interventions: Dietary Supplement: Alpha Lipoic Acid Supplement
- Cellulose Fiber Placebo (Placebo Comparator): 600mg/daily ingestion of Vital Nutrients placebo (cellulose starch) with no change in lifestyle for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid Supplement — Alpha lipoic acid ingestion (600mg/daily) for 8 weeks with no change in lifestyle.
  Arms: GNC Alpha Lipoic Acid Supplement
Dietary Supplement: Placebo — Cellulose fiber ingestion (600mg/daily) for 8 weeks with no change in lifestyle.
  Arms: Cellulose Fiber Placebo

SUMMARY:
Eight weeks supplementation of alpha lipoic acid (known superantioxidant already produced by the body) will significantly improve metabolic syndrome markers (e.g., excess body weight, blood pressure, glucose, insulin, blood lipids, and self-report measures) in young (18-25 years) overweight or obese males compared to placebo (cellulose starch). If the hypothesis is supported, alpha lipoic acid ingestion could be beneficial in reducing disease risk and enhancing metabolic dysfunction in ethnic individuals. Therefore, the purpose is to establish the impact alpha lipoic acid has on the modifiable markers associated with metabolic perturbations consistent with metabolic syndrome in males.

DETAILED DESCRIPTION:
Young adults exhibit an increasing prevalence of obesity, pre-diabetes, and metabolic syndrome that contribute to increased risk of type II diabetes and cardiovascular heart disease later in life. Twenty five percent of American adults have been diagnosed with metabolic syndrome, whereas the prevalence increases to 30 % in Mexican American adults between 30-70 years old. The risk in this population may be higher based on ethnicity and the rising obesity rates in young adults and children, although the definition of metabolic syndrome in younger age has yet to be established. Factors causing metabolic syndrome are complex but include a physically inactive lifestyle, an unhealthy diet made up of saturated fat and processed foods, and inherited influences. Therefore identifying the need to intervene early with a dietary intervention in order to combat the risk for future disease is vital. It is hypothesized that 8 weeks supplementation of alpha lipoic acid (known superantioxidant already produced by the body) will significantly improve metabolic syndrome markers (e.g., excess body weight, blood pressure, glucose, insulin, blood lipids, and self-report measures) in young (18-25 years) overweight or obese males compared to placebo (cellulose starch). If the hypothesis is supported, alpha lipoic acid ingestion could be beneficial in reducing disease risk and enhancing metabolic dysfunction in young individuals. Therefore, the purpose is to establish the impact alpha lipoic acid has on the modifiable markers associated with metabolic perturbations consistent with metabolic syndrome in males.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (body mass index 25 - 35 kg/m2)
* Males (18-35 years)
* Able to ingest supplement or placebo

Exclusion Criteria:

* Female (due to menstrual cycle fluctuations)
* Unable to read English at the time of consent
* Have a body mass index under 25 kg/m2 or over 35 kg/m2
* Diabetes
* Impaired glucose tolerance (fasting plasma glucose levels >110 mg/dL
* Hypertension (SBP>130mmHg or DBP>90mmHg)
* Cardiovascular problems or disease
* Psychiatric problems
* History of alcohol abuse (intake of >500 g/wk in the last year)
* Current or recent (in the past 3 years) smoking
* Certain medication or dietary supplement use (medications or dietary supplements known to cause weight loss/gain or metabolic improvements/dysfunction. Paxil or (paroxetine), Prozac (fluoxetine), Remeron (mirtazapine), Zyprexa (olanzapine), Deltasone (prednisone), Thorazine (chlorpromazine), Elavil, Endep, Vanatrip (amitriptyline), Depakote (valproic acid), Allegra (fexofenadine and pseudoephedrine), Diabinese or Insulase
* Symptoms of chronic or current infection
* A chronic inflammatory condition
* Any thyroid condition, and/or liver disease or malignancy

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Effects on whole blood fasting glucose | 8 weeks
  Measured by single drop cuvette of whole blood using Hemocue Glucose 201
Effects on fasting plasma inflammatory biomarkers | 8 weeks
  Measured by ELISA kit
Effects on body composition (body fat, muscle mass, body weight) | 8 weeks
  Measured by bioelectrical impedance using a Tanita floor scale

SECONDARY OUTCOMES:
Effects on oxygen consumption and carbon dioxide production at rest | 8 weeks
  Measured by True One Metabolic Cart by Parvomedics via hood
Effects on oxygen consumption and carbon dioxide production during exercise | 8 weeks
  Measured by True One Metabolic Cart by Parvomedics via facemask

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Dunn, Ph.D., Principal Investigator — University of La Verne Assistant Professor
Locations (1):
- University of La Verne Kinesiology Laboratory, La Verne, California, United States

IPD SHARING:
Plan to Share IPD: Undecided